CLINICAL TRIAL: NCT02205450
Title: Experience With Growth Hormone (GH) in Children Under 2 Years With Prader-Willi Syndrome (PWS) in the Pediatric Endocrine Department of the Hospital of Sabadell
Brief Title: Growth Hormone in Children Under 2 Years With Prader-Willi in Hospital of Sabadell
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Raquel Corripio-Collado, MD PhD, Corporacion Parc Tauli
Other Study IDs: CPT_ENDOPED201401
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; Growth Hormone; Children
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children under 2 years with Prader-Willi Syndrome
  Interventions: Drug: Recombinant Somatropin

INTERVENTIONS:
Drug: Recombinant Somatropin

SUMMARY:
The PWS is a genetic disease with intellectual disabilities associated with multiple manifestations in other body systems. It is characterized by hypothalamic-pituitary abnormalities with severe hypotonia during the early years of life, conditioning feeding difficulties. Hyperphagia appears later, causing severe obesity in pre - school ages. Other endocrine abnormalities associated produce short stature, GH deficiency and hypogonadotropic hypogonadism. These patients also have varying cognitive dysfunction associated as well as learning problems, compounded by the development of psychological-psychiatric and behavioral problems language. The aetiology of GH decreased secretion of the SPW is controversial, it is known that IGF -1 levels are reduced in children and adults with PWS. The rational use of GH is derived from knowledge of comorbidities observed in PWS, which seem to be related to GH deficiency: hypotonia, altered body composition, decreased growth, even obesity.

• The GH is accepted since 2000 for the treatment of PWS. Following fatal episodes in our country, it was decided to start treatment at 2 years of age in an arbitrary manner, but not in the U.S. or France. Subsequent studies have found that GH per se is not a risk factor for mortality. The currently published data supporting the benefits of GH treatment when started between 4 and 6 months of life, even some experts advocate starting at 3 months, but due to the lack of consensus on the age of onset treatment, despite the benefits of your home at an early age before the onset of obesity often starts around 2 years of life.

HYPOTHESIS The use of GH is safe and effective in patients with PWS children under 2 years old.

ELIGIBILITY:
Inclusion Criteria:

* Children under 2 years

Exclusion Criteria:

-

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalary population
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
To assess the safe use of GH in children under 2 year old with Prader Willi Syndrome | Two years
  Collect any Serious Adverse Event during the length of study

SECONDARY OUTCOMES:
Evaluate the impact of treatment with GH in kids under 2 years old on body composition | Every 3 months during 2 years
Evaluate the impact of treatment with GH in kids under 2 years old on start walking | Every 3 months during 2 years
Evaluate the impact of treatment with GH in kids under 2 years old on the speech beginning | Every 3 months during 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Corripio, PI, Principal Investigator — Corporacio PT
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- See also: Safety and effectiveness of growth hormone therapy in infants with Prader-Willi syndrome younger than 2 years: a prospective study Raquel Corripio ORCID logo, Carla Tubau, Laura Calvo, Carme Brun, Núria Capdevila, Helena Larramona and Elisabeth Gabau — https://doi.org/10.1515/jpem-2018-0539